CLINICAL TRIAL: NCT04573413
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation (r-TMS) Combined With Visual Scanning Treatment on Cognitive-behavioral Symptoms of Unilateral Spatial Neglect in Patients With Traumatic Brain Injury: a Randomized Clinical Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation in Traumatic Brain Injury
Acronym: Smart trace
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Fabio La Porta (Unknown); Francesco Di Gregorio (Unknown); Roberto Piperno (Unknown); Emanuela Casanova (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SG-2018-12367527
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Perceptual Disorders; Traumatic Brain Injury
Keywords: Electroenephalography; repetitive Transcranial magnetic stimulation; Hemispatial Neglect
MeSH Terms: conditions — Perceptual Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- r-TMS group (Experimental): The interventions have a total administration time of 75 minutes per day. For rTMS stimulation, the coil will be positioned tangentially on the target area. Each rTMS session will last 15 minutes and will be administered every other day (e.g. Monday-Wednesday-Friday, Monday-Wednesday-Friday, Monday). The CCT (i.e. visual scanning treatment) involves the presence of a therapist, who administers various visual scanning tasks, used to increase patient's awareness and to teach strategies to improve spatial exploration abilities.Trainings include three increasing levels of difficulty (9 possible combinations). Each level of difficulty will be exercised until the patient reaches a level of accuracy of 75%. The CCT will be carried out in 50 minutes sessions for 5 days a week within 15 days (11 sessions in total). On the days when the rTMS is also administered, the administration of the CCT will immediately follow the brain stimulation.
  Interventions: Device: Inhibitory repetitive transcranial magnetic stimulation
- SHAM group (Sham Comparator): SHAM Stimulation and Visual Scanning training. In the control group, the coil of the r-TMS will be positioned at 90° on the target area, thus no specific cortical modulation will be implemented (SHAM stimulation). For the SHAM group, the CCT protocol will be administered with the same modalities and time frame as detailed for the experimental group.
  Interventions: Device: Sham Group

INTERVENTIONS:
Device: Inhibitory repetitive transcranial magnetic stimulation — r-TMS Parameters: International 10/20 system for the location of the target area (left parietal cortex) 60% Power Frequency: 1 Hz 90 pulse trains with 10 pulses each (total 900 stimuli), resulted in a total stimulation period of 15 minutes.
  Visual Scanning Visual-spatial training; Reading and copying training; Copying of line drawings on a dot matrix. Barrage
  Arms: r-TMS group
Device: Sham Group — Sham stimulation and Visual scanning training Intervention: Device: SHAM
  Arms: SHAM group

SUMMARY:
Randomized Controlled Trial (RCT) aiming at assessing the efficacy of a novel rehabilitation protocol, based on repetitive transcranial magnetic stimulation (r- TMS) in combination with a conventional cognitive treatment (CCT). The protocol will be statistically compared to the same CTT administered without the r-TMS in a sample of traumatic brain injury patients (age between 18 and 80 years) with left hemispatial Neglect.

DETAILED DESCRIPTION:
BACKGROUND: A frequent and disabling impairment in persons who suffered traumatic brain injury (TBI) is left hemi-spatial neglect (LHSN). LHSN is a spatial attentive syndrome, characterized by a reduced ability to attend, perceive and consciously represent the left contra-lesional space, in the absence of a primary sensory deficit. Persons with LHSN fail to attend any stimulus coming from the left space and this can affect the ability to carry out many everyday tasks, such as walking, eating, reading and getting dressed. Those patients, as a direct consequence of the brain injury and LHSN, are also often affected by anosognosia for hemiplegia and for LHSN, which is the lack of awareness about motor and cognitive deficits. This condition hinders motor and cognitive recovery, predisposes to falls and reduces independence. Furthermore, in TBI LHSN is often associated with a mixture of attention, memory, executive function, and processing speed deficits leading to complex cognitive and behavioral pictures, which may even interfere with the administration of standard cognitive treatments for LHSN (i.e. visual scanning protocols or prism adaptation). It is also known that 1 Hz inhibitory repetitive Transcranial Magnetic Stimulation (rTMS), applied for two weeks to the posterior parietal cortex (PPC) of the unaffected hemisphere in patients with LHSN due to ischemic lesion of the right hemisphere, induces a significant improvement of visual-spatial symptoms that persists 15 days after rTMS treatment. These results can be explained considering that spatial attention deficit in LHSN due to a right middle cerebral artery territory stroke relates to abnormal activation of neural system that mediates spatial attentive operations in the healthy brain. In LHSN, a lesion of the right PPC and of the inter-hemispheric connectivity causes an imbalance in interhemispheric activity due to hyperactivity of the left hemisphere which, in turn, causes a biased attentive allocation towards ipsilesional space. As a consequence, an inhibition of this hyperactivity may have a rebalancing effect, reducing left spatial attention deficit in LHSN. Indeed, recent studies in stroke showed also the possibility of improving the efficacy of standard cognitive treatments (i.e. visual scanning) if the latter are preceded by inhibitory rTMS on the unaffected hemisphere. What is not known is whether also in LHSN due to TBI, inhibitory rTMS on the left PPC followed by a visual scanning protocol may be an effective treatment as in right hemisphere stroke, considering that in TBI the damage is often more widespread and multifocal than in the former condition.

AIMS:

* To compare the efficacy of a combined r-TMS and CCT intervention aiming at reducing cognitive symptoms of LHSN, in a sample of TBI patients with LHSN, within the context of an RCT.
* To evaluate the long- term impact of the intervention and evaluate the effect of the intervention on several clinical measures (activity of daily living, attentive and motor functions) and on psychophysiological indices

METHODS: Randomized controller trial, with blind assessments on pretest, postest and on 3 months follow-up.

POPULATION: TBI patients with clinical evidence of LHSN. INTERVENTION: Inhibitory low-frequency r-TMS on the left parietal cortex combined with a conventional cognitive treatment (visual scanning training) for 2 weeks.

CONTROL: SHAM group with a placebo r-TMS stimulation combined with visual scanning training for 2 weeks.

OUTCOMES: Multidisciplinary assessment with clinical and psychophysiological indices. The primary endpoint is a psychophysiological index based on Visual-Evoked Potentials (VEPs). In particular we will focus on the N1 component, a posterior negativity, which is altered in terms of latency and amplitude in LHSN population. In order to study effects of the r-TMS in the interhemispheric parietal pathway, we will extract indices of interhemispheric transmission time (IHTT) on the N1 latency and of spatial attention bias on N1 amplitude (VABI). The secondary outcomes will consider the impact of the intervention on other clinical measures of cognitive and motor impairment and on test of activity of daily living.

EXPECTED RESULTS: The main expected outcome of the present project will provide evidence, on a large simple of TBI patients, of the interhemispheric functionality underlying cognitive symptoms of LHSN. It will point out the specific effect of rTMS protocols on the inter-hemispheric imbalance. More in details, we expect to observe in the rTMS group a larger rebalancing effect than in the control group, as demonstrated by psychophysiological indexes, with the persistence of effects at follow-up. Additionally, we expect to observe larger improvements in cognitive and behavioral symptoms of LHSN induced by the rTMS in comparison to the control group, as demonstrated by better performances on clinical tests and batteries.

RANDOMIZATION: In order to ensure that each arm will contain an equal number of individuals, eligible subjects will be randomly assigned to one of the two groups with a blocked randomization method based on a block size of 4.

ASSESSOR AND PATIENT BLINDNESS: In order to ensure a double-blind assessment, pre-treatment assessments will be performed prior to randomization. An assessor not aware of the patient randomization group will conduct post-treatment and follow-up assessments. Also the visual scanning protocol will be administered by therapists unaware of the patient randomization and patients themselves will be instructed not to reveal any information on the brain stimulation treatment received.

CASE REPORT AND DATA MONITORING: Specific case report forms (CRF) for every test in the assessments are already available and will be used. During the treatment the responsible physician will report any adverse event in the treatment-CRF. All information and results will be promptly reported on the electronic database. A researcher will be responsible for the electronic database, data analyses and will draft the single patient record at the end of all procedures. In case of lost to follow-up, the information available up to that moment will be considered. If participant is lost at follow-up, it will be analyzed on the basis of the "intention to treat" principle. Finally, the reason for quit the study will be reported for each participant lost at follow-up.

SAMPLE SIZE: The sample size was calculated using the following formula:

https://www.dropbox.com/s/y56umrt7z93en1w/Simple%20size%20formula.docx? dl=0 The sample size resulting from the formula calculated for the VABI is 24. Consequently, the minimum sufficient sample to reach the primary aim is, assuming approximately 10% of subjects lost to follow-up, 28 subjects (14 X group) recruited over a three-year period.

DATA ANALYSES: Analysis of covariance will be performed for each measure using a mixed-model ANCOVA with a 2X3 design, where the "between" factor is represented by the randomization groups (rTMS, SHAM) and the "within" factor is the assessment time (T0, T1, T2). Data analysis will be performed using Matlab and SPSS softwares.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of TBI;
2. Diagnosis of LHSN with specific assessment tests (line bisection test and / or star cancellation test);
3. Intra-hospital rehabilitation setting (ordinary hospitalization or DH);
4. Age between 18 and 80 years;
5. Time after injury between three weeks and 1 year;
6. Level of cognitive functioning (LCF ≥5 )
7. Adequate language comprehension

Exclusion Criteria:

1. Clinical instability at enrollment (for example, fever, acute internist conditions, etc.);
2. Presence of epileptogenic alterations to the EEG and / or previous epileptic seizures;
3. Presence of intracranial implants of metallic material;
4. Presence of devices that could be altered by rTMS, such as pacemakers, ventriculo-peritoneal derivations, Baclofen pump;
5. Acute neurosurgery, including decompressive craniotomy;
6. Drugs conditioning the state of consciousness-vigilance such as benzodiazepines;
7. Cortical blindness and / or visual agnosia;
8. Concomitant psychiatric disorders and / or history of substance abuse;
9. Post-traumatic agitation
10. Post-traumatic complications (i.e. hydrocephalus)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
visual-Attention Bias Index (vABI) | up to 21 days post baseline and up to 90 days follow-up
  Change from Baseline: visual-Attention Bias Index (vABI). Psychophysiological index of inter-hemispheric imbalance in a visual-spatial attention task

SECONDARY OUTCOMES:
behavioral Inattention Test (BIT) | up to 21 days post baseline and up to 90 days follow-up
  1. Change from Baseline: behavioral Inattention Test (BIT). A battery for the assessment of cognitive and behavioral symptoms in LHSN
catherine Bergegò Scale (CBS) | up to 21 days post baseline and up to 90 days follow-up
  2. Change from Baseline: catherine Bergegò Scale (CBS). A battery for the assessment of LHSN symptoms in the activity of daily living.
test of Attention Performance (TAP/TEA) | up to 21 days post baseline and up to 90 days follow-up
  3. Change from Baseline: test of Attention Performance (TAP/TEA). Two subtest will be executed "alertness" and "Visual field/Neglect" to assess attentive functions
functional independence measure (FIM) | up to 21 days post baseline and up to 90 days follow-up
  4. Change from Baseline: functional independence measure (FIM). The motor subscale will be executed to assess motor independence
Motricity Index (MI) | up to 21 days post baseline and up to 90 days follow-up
  5. Change from Baseline: Motricity Index (MI). A test to assess motor impairment in stroke patients
Trunk Control Test (TCT) | up to 21 days post baseline and up to 90 days follow-up
  6. Change from Baseline: Trunk Control Test (TCT). A test to assess the ability to control the trunk after stroke.
Inter Hemispheric transmission Time (IHTT) | up to 21 days post baseline and up to 90 days follow-up
  7. Change from Baseline: Inter Hemispheric transmission Time (IHTT). Psychophysiological index of inter-hemispheric transmission time.
Level of Cognitive Functioning (LCF) | up to 21 days post baseline and up to 90 days follow-up
  8. Change from Baseline: Level of Cognitive Functioning (LCF). A test to assess general cognitive functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Unità Sanitaria Locale di Bologna 40124, Bologna, Italy, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Gregorio F, La Porta F, Lullini G, Casanova E, Petrone V, Simoncini L, Ferrucci E, Piperno R. Efficacy of Repetitive Transcranial Magnetic Stimulation Combined With Visual Scanning Treatment on Cognitive-Behavioral Symptoms of Unilateral Spatial Neglect in Patients With Traumatic Brain Injury: Study Protocol for a Randomized Controlled Trial. Front Neurol. 2021 Jul 14;12:702649. doi: 10.3389/fneur.2021.702649. eCollection 2021. PMID 34335455
- See also: Related Info — http://doi.org/10.1007/s10072-013-1412-y